CLINICAL TRIAL: NCT03059953
Title: A Non-interventional, Prospective, Observational Study of Treatment With APRemilast in Moderate psoriAsIS in Real Life clinicAL Practice (The 'APRAISAL' Study)
Brief Title: A Study of Treatment With APRemilast in Moderate psoriAsIS in Real Life clinicAL Practice (The 'APRAISAL' Study)
Acronym: APRAISAL
Status: Completed | Type: Observational
Sponsor: Genesis Pharma S.A. (Industry)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: GEN-NIS-APR-001
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-05

CONDITIONS: Moderate Plaque Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
For patients with moderate plaque psoriasis who are intolerable to, have a contraindication to or have failed classical systemic treatments, the current commonly employed management strategy encompasses treatment with biologic agents. The direct and indirect costs of biologic treatment, accruing, among others, from the high drug acquisition and administration costs, the required baseline safety screening and subsequent routine monitoring as well as the potential loss of patients' working hours constitute a significant financial burden on the public healthcare system. In light of the above evidence, it appears that in routine care apremilast may fulfill an important gap in the treatment armamentarium of psoriasis by providing a promising treatment option to be employed prior to biologics, which has demonstrated efficacy even in hard-to-treat areas such as the scalp, nails, palms and soles, and has a limited manageable safety profile, while being more convenient and cost-effective than biologics.

In view of the scarcity of real-world evidence regarding the impact of apremilast on the patients' health-related quality of life (HRQoL) and extent and severity of the disease, and under the consideration that the moderate psoriasis patient {defined as [10<body surface area (BSA)<20 or 10<psoriasis area severity index (PASI)<20] and 10<dermatology quality of life index (DLQI)<20}, naïve to biologic treatment was likely underrepresented in the pivotal ESTEEM trials since approximately 30% of the enrolled patients had been previously treated with biologic therapy, 28-30% had a baseline PASI score >20, and 48-52% had a BSA >20%, this study represents an attempt to examine the impact of apremilast in routine clinical practice settings in Greece on the patient with moderate plaque psoriasis when this therapeutic strategy precedes biologics in the treatment algorithm.

Specifically, the present study aims to generate novel real-world evidence on the effect of apremilast treatment in biologic treatment naïve patients with moderate plaque psoriasis in terms of the patients' HRQoL, patient-perceived benefits of therapy, treatment response rate, and impact on nail, scalp and palmoplantar psoriatic involvement and severity of pruritus, while concurrently assessing apremilast survival rate and cost per PASI-75 responder in the routine clinical practice of Greece.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study have to meet all of the following criteria:

* Male and female patients ≥ 18 years of age at the time of informed consent;
* Patients diagnosed with moderate chronic plaque psoriasis [(10<BSA<20 or 10<PASI<20) and 10<DLQI<20], who failed to respond to or who have a contraindication to, or are intolerant to other classical systemic therapy;
* Patients naïve to biologic treatments;
* Patients for whom the decision to prescribe therapy with apremilast (Otezla®) according to the locally approved summary of product characteristics (SmPC) has already been taken prior to their enrollment in the study and is clearly separated from the physician's decision to include the patient in the current study;
* Patients with available BSA, PASI and DLQI scores at the start of apremilast treatment;
* Patients must be able to read, understand and complete the study specific questionnaires;
* Patients must provide a written Informed Consent prior to inclusion to the study;
* Patients must be able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from participation in this study:

* Patients who have initiated treatment with apremilast more than 7 days before enrollment into the study;
* Patients that meet any of the contraindications to the administration of the apremilast as outlined in the latest version of the locally approved SmPC;
* Patients currently receive treatment with any investigational drug/device/intervention or who have received any investigational product within 30 days or 5 half-lives of the investigational agent (whichever is longer) before the commencement of therapy with apremilast;
* Patients who are currently pregnant, breastfeeding, or planning a pregnancy during the study observation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients ≥ 18 years of age, diagnosed with moderate chronic plaque psoriasis [(10<BSA<20 or 10<PASI<20) and 10<DLQI<20], who failed to respond to or who have a contraindication to, or are intolerant to other classical systemic therapy and naïve to biologic treatments
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Quality of Life - Percentage of patients with moderate plaque psoriasis treated with apremilast who will achieve a DLQI total score ≤ 5 (i.e., no or small effect of their skin problem on HRQoL) | at 24 weeks post-treatment onset
  Percentage of patients with moderate plaque psoriasis treated with apremilast who will achieve a DLQI total score ≤ 5 (i.e., no or small effect of their skin problem on HRQoL)

CONTACTS AND LOCATIONS:
Locations (1):
- 401 General Military Hospital, Athens, Greece

REFERENCES:
- [Result] Ioannides D, Antonakopoulos N, Georgiou S, Chasapi V, Katsantonis I, Drosos A, Rigopoulos D, Antoniou C, Anastasiadis G, Bassukas I, Ioannidou D, Protopapa A, Neofotistou O, Krasagakis K, Aronis P, Papageorgiou M, Lazaridou E, Patsatsi A, Lefaki I, Roussaki-Schulze AV, Satra F, Anagnostopoulos Z, Papakonstantis M. Effectiveness and safety of apremilast in biologic-naive patients with moderate psoriasis treated in routine clinical practice in Greece: the APRAISAL study. J Eur Acad Dermatol Venereol. 2021 Sep;35(9):1838-1848. doi: 10.1111/jdv.17392. Epub 2021 Jul 13. PMID 34036627